CLINICAL TRIAL: NCT04605263
Title: Effects of Deep Brain Stimulation (DBS) of the Pedunculopontine Nucleus (PPN) on Gait, Postural Stability, Freezing of Gait (FOG), and Falls
Brief Title: Deep Brain Stimulation (DBS) of the Pedunculopontine Nucleus (PPN)
Acronym: PPNGB01
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: St. Joseph's Hospital and Medical Center, Phoenix (Other)
Collaborators: Arizona State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: PHX-19-500-412-30-04
Record Dates: First submitted 2020-08-31; First posted 2020-10-27 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Parkinson Disease
Keywords: Deep Brain Simulation (DBS); Gait and Balance; Postural Instability and Gait Dysfunction (PIGD)
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Patients will be randomly assigned (1:1) to receive either traditional STN stimulation or STN+PPN patients. Once implanted, all patients will receive stimulation of all implanted devices for the first three months to allow for stimulation parameters to be adjusted. During this time, STN+PPN subjects will have their PPN stimulation parameters mapped (all DBS contacts in the PPN will be tested to determine which stimulation pattern achieves best results). Once patients have been tested at the 3-month post-op visit, STN+PPN patients will be double-blindly randomized (1:1) to either receive or not receive PPN stimulation for the following six months before further testing. Following the 9-month testing visit, STN+PPN patients will be crossed over so that those receiving PPN stimulation before will have their device turned off, and vice versa. After further testing at 15 months, all patients will have their devices turned back on. There will be one final test at 27 months.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- STN DBS (Active Comparator): Subjects will receive traditional bilateral STN devices and stimulation.
  Interventions: Procedure: Deep Brain Stimulation Surgery (DBS)
- STN-PPN DBS (Experimental): Patients will be implanted with both bilateral STN and bilateral PPN devices. These patients will undergo a crossover between 3 and 15 months post-op in which they will double-blindly receive PPN stimulation for six months and have stimulation turned off for six months. All patients will receive stimulation from 0-3 months post-op (mapping visits occur in this window) and from 15-27 months.
  Interventions: Device: STN-PPN DBS Surgery

INTERVENTIONS:
Device: STN-PPN DBS Surgery — Subject will undergo standard bilateral STN DBS surgery and have 2 additional leads placed in the same burr with bilateral PPN targets
  Arms: STN-PPN DBS
Procedure: Deep Brain Stimulation Surgery (DBS) — DBS lead implantation of bilateral STN
  Arms: STN DBS

SUMMARY:
This is a mechanistic study to determine the differential effects of the dopaminergic and cholinergic systems on attention, gait, and balance. The primary goal of the study is to evaluate the relative effects of pedunculopontine nucleus (PPN) and subthalamic nucleus (STN) Deep Brain Stimulation (DBS) on these features in persons with Parkinson's Disease (PD) who are eligible for DBS for improvement of their motor symptoms and exhibit gait instability with falls. Patients will be enrolled and implanted with bilateral electrodes in one of the approved DBS locations (subthalamic nucleus: STN), but additionally electrodes will be inserted into the experimental target, namely the PPN bilaterally.

DETAILED DESCRIPTION:
This is a prospective, single-center randomized controlled trial designed to estimate the potential clinical benefit, and associated risks, of deep brain stimulation of the of the PPN and STN in patients with PD that are candidates for DBS for improvement of their motor symptoms and exhibit gait instability with falls. Patients will be enrolled and implanted with additional bilateral electrodes in the PPN. Each subject will be randomized 1:1 to one of the following sequences: Bilateral STN+PPN stimulation or Bilateral STN stimulation alone. The addition of a bilateral STN stimulation only group allows for the research of potential micro-lesioning effects of the PPN which might affect features of interest even in the absence of PPN stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria

  1. Informed consent signed by the subject.
  2. Diagnosed with Parkinson's disease per UK Parkinson's Disease Society Brain Bank (Queens Square) criteria for at least 4 years
  3. Demonstrates levodopa responsiveness of at least 30%
  4. Experiences tremor or motor complications including wearing off and/or dyskinesia
  5. DBS candidate per FDA guidelines as outlined in criteria 2-4
  6. Candidate for STN targeting per the consensus committee
  7. Subject exhibits gait instability, or a history of at least one fall within the last year, or a history of falls on tests of Static or Dynamic Stability.
  8. PD Stage 2-3 with predominant axial symptoms or FOG refractory to Levodopa > 600 mg and UPDRS Part III Subscore of >6.
  9. Subject is ambulatory and able to walk for limited periods of time without using an assistive device.
  10. 18-75 years of age
  11. Primary English speaking
  12. Physically and cognitively capable of completing evaluations and consent
  13. Medically cleared for surgery and anesthesia
  14. Female subjects with child-bearing potential have a negative serum pregnancy test prior to DBS surgery

Exclusion Criteria:

Exclusion Criteria:

1. Dementia per DSM-V criteria
2. Condition precluding MRI
3. History of supraspinal CNS disease other than PD
4. History of schizophrenia, delusions, or currently uncontrolled visual hallucinations
5. Subjects who require rTMS, ECT, diathermy, or repeat MRI procedures to treat a medical condition.
6. Subjects with a history of seizure disorder
7. Subjects who have made a suicide attempt within the prior year,
8. Subjects with any medical contraindications to undergoing DBS surgery (eg, infection, coagulopathy, or significant cardiac or other medical risk factors for surgery)
9. Subjects with an implanted stimulator such as a cardiac pacemaker, defibrillator, neurostimulator and cochlear implant
10. Subjects who are pregnant or nursing.
11. Patient that is unwilling or unable to comply with the requirements of this protocol, including the presence of any condition (physical, mental, or social) that is likely to affect the subject's ability to comply with the protocol.
12. Any other reasons that, in the opinion of the investigator, the candidate is determined to be unsuitable for entry into the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
STN-PPN Stimulation Effect on Fall Risk | 27 months
  The purpose of this study is to measure the effect and the mechanism of deep brain stimulation (DBS) of the pedunculopontine nucleus (PPN) on fall risk as established by quantitative gait and balance analysis.

SECONDARY OUTCOMES:
STN-PPN on Linear and Nonlinear Measures of Gait | 27 months
  Linear and nonlinear measured of gait will be measured during straight walking, turning, and arising and returning to a chair.
STN-PPN on Linear and Nonlinear Measures of Balance | 27 months
  Linear and nonlinear measures of balance will be collected during eyes open, eyes closed, and perturbed (dyanic balance) conditions.
STN-PPN on Attention | 27 months
  The effect of PPN stimulation, in comparison to that of STN alone, on attention, with be measured using the Conners Continuous Auditory Test of Attention and Continuous Performance Test 3.
STN-PPN on Subjective Measures of Alertness | 27 months
  The effects of PPN stimulation on subjective function will be measured using the Toronto Alertness Scale, graded 0-50, with higher scores being better.
STN-PPN on Subjective Measures of Sleep | 27 months
  The effects of PPN stimulation on subjective function will be measured using the Epworth Sleep Scale, graded 0-24, with lower scores being better.
STN-PPN on Subjective Measures of Non-Motor Symptoms | 27 months
  The effects of PPN stimulation on subjective function will be measured using the Non-Motor Symptom Assessment, graded 0-360, with lower scores being better.
STN-PPN on Subjective Measures of Balance in Daily Life | 27 months
  The effects of PPN stimulation on subjective function will be measured using the Activity-specific Balance Confidence Scale, graded on a scale of 0-100, with higher scores being better.

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Moguel-Cobos, MD, Principal Investigator — Muhammad Ali Movement Disorders Clinic Physician
Locations (1):
- St. Joseph's Hospital & Medical Center / Barrow Neurological Institute, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No
There is a Data Use Agreement (DUA), with Boston Scientific.